CLINICAL TRIAL: NCT05684198
Title: Emergency Laparotomy for Peritonitis and Surgical Site Infection: Preventive Subcutaneous NPWT vs Primary Closure - a Randomized Health Services Study
Brief Title: NPWT vs Primary Closure in SSI Prevention for Emergency Laparotomies for Peritonitis
Acronym: PRISTINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 420/1
Record Dates: First submitted 2022-11-29; First posted 2023-01-13 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2023-05

CONDITIONS: Peritonitis; Surgical Site Infection; Infections; Wound Infection
Keywords: laparotomy; NPWT; primary closure; vacuum-assisted closure; VAC
MeSH Terms: conditions — Peritonitis; Surgical Wound Infection; Infections; Wound Infection | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- subcutaneous NPWT (Experimental): The peritoneum and fascia will be closed as in the PC arm. Subsequently, patients will be treated with commercially available vacuum-assisted closure systems (provided by Smith&Nephew or Hartmann) according to the manufacturer's instructions. Following fascia closure, the NPWT foam will be adjusted to the wound size to fill the wound cavity without causing excessive wound dehiscence. Subsequently, the foam will be placed in the subcutaneous tissue. The foam will not be fixated on the skin with sutures. The wound will be sealed with adhesive film. In case of air leak in problematic areas such as the navel or ostomy, ostomy paste will be used to create a tighter seal. Continuous pressure of 120 mmHg will be applied. On the 3rd day postop, the dressing will be removed and closure by secondary intention will be performed.
  Interventions: Device: subcutaneous NPWT
- primary closure (No Intervention): The peritoneum will be closed as a separate layer with a 2-0 multifilament absorbable suture. Subsequently, the fascia will be closed with a continuous suture using absorbable monofilament 0 sutures. Subcutaneous tissue will be rinsed twice with hypochlorite solution following peritoneal closure and fascial closure. Interrupted subcutaneous closure will be performed with absorbable multifilament 2-0 sutures. Following skin disinfection with an alcohol solution, the skin will be closed with non-absorbable monofilament 2-0 or 3-0 sutures using the interrupted mattress technique. Conventional Cosmopor® sterile gauze dressings will be applied. Unless the dressing material will be saturated, the dressing will remain unchanged until 3rd day post-op.

INTERVENTIONS:
Device: subcutaneous NPWT — Following fascia closure, NPWT system will be inserted into subcutaneous tissue, continuous negative pressure of 120 mmHg will be applied.
  Other Names: vacuum-assisted wound closure; Vivano; Renasys
  Arms: subcutaneous NPWT

SUMMARY:
The study aims to evaluate the efficacy of negative pressure wound therapy (NPWT) compared with primary closure (PC) in surgical site infection (SSI) prevention for laparotomy for peritonitis.

DETAILED DESCRIPTION:
Surgical site infection is a particularly common morbidity in contaminated surgeries leading to prolonged length of hospital stay, healing time, and a significant financial burden on healthcare systems.

Hence, the objective of PRISTINE trial is to compare the effectiveness of subcutaneous NPWT with PC for SSI prevention in patients who, due to wound contamination, are prone to infection. Moreover, with a further cost analysis, the investigators aim to evaluate the rationale for the implementation of routine preventive NPWT for laparotomy for diffuse peritonitis.

Patients qualified for an emergency laparotomy for peritonitis in University Clinical Centre (UCC) Division of Oncological, Endocrine and General Surgery will be identified. Prior to laparotomy, participants will be randomized in 1:1 ratio to subcutaneous NPWT or PC. The assigned intervention will be performed intraoperatively, after fascia closure.

All participants will receive an empirical antibiotic therapy regimen consisting of tazobactam/piperacillin or ciprofloxacin+ metronidazole. Participants will be followed-up postoperatively for one year.

In case of an SSI all participants, regardless of their initial allocation, will be treated according to the standard of care with prolonged NPWT and targeted antibiotic therapy.

ELIGIBILITY:
Inclusion Criteria:

* qualified for an emergency laparotomy for peritonitis
* gave written informed consent

Exclusion Criteria:

* qualified for open abdomen treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-01-11 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Effective wound closure by 30th day post-op | 30 days
  definitive wound closure, not followed by secondary wound dehiscence
Time to end of surgical treatment of the wound | 1 year
  Time of last out-patient visit ending the process of treating surgical wound

SECONDARY OUTCOMES:
Length of stay | 90 days
  postoperative length of hospital stay
Time to heal | 120 days
  time to full epithelialisation of the wound
Volume of wound drainage | 60 days
  Volume of wound drainage collected in a NPWT or drainage collector
Time of secondary NPWT treatment | 60 days
  Duration of NPWT therapy administered if SSI occured
Post-operative morbidity | 60 days
  occurrence of adverse events and complications following surgery measured with Clavien-Dindo scale (grade I to V; grade I represents any deviation from the normal post-operative course not requiring surgical, endoscopic or radiological intervention and grade 5 represents patient's death)
SSI presence or absence | 30 days
  Surgical Site Infection according to Centre for Disease Control (CDC) criteria:
  Infection occurring within the first 30 post-operative days with at least one of the following:
  * Purulent drainage from the incision
  * Organisms isolated from an aseptically obtained culture of fluid or tissue from the incision
  * Incision is deliberately opened by a surgeon AND at least one of the following signs/symptoms of infection:
    1. Pain or tenderness
    2. Localized swelling
    3. Redness
    4. Heat
  * Diagnosis of SSI by the surgeon or attending physician
  Due to the inability to implement CDC for wounds treated with NPWT, the investigators have included additional SSI criteria: the absolute necessity to prolong NPWT after 3rd day postop, an anergic wound morphology or slough.
Pain level | 7 days
  Pain measured with Visual Analogue Scale every 8h (subjective pain strength scale from 0 to 10; 0 represents no pain and 10 represents the worst pain)
Scar quality | 1 year
  Measured with Vancouver Scar Scale (VSS). This scale ranges from 0 (representing normal skin) to 13 (representing worst scar imaginable). VSS provides the assessment of the following wound characteristics: pigmentation (0-2), vascularity (0-3), pliability (0-5), height (0-3).
Cost | 1 year
  Cost of hospitalisation and outpatient visits

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Spychalski, MD PhD, Principal Investigator — MUG Division of General Surgery; Katarzyna M Polomska, Principal Investigator — Medical University of Gdansk (MUG); Jaroslaw Kobiela, Prof., Principal Investigator — MUG Division of General Surgery
Locations (1):
- UCC Division of Oncological, Transplant and General Surgery, Gdansk, Pomeranian Voivodeship, Poland